CLINICAL TRIAL: NCT00888407
Title: Community-based Hepatitis B Interventions for Hmong Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200614458; P01CA109091 (NIH)
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-12

CONDITIONS: Liver Cancer
Keywords: Asian American Health; Cancer; Hepatitis; Hepatitis B; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Hepatitis; Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBV Screening (Experimental): Small group educational session with HBV screening resources provided.
  Interventions: Behavioral: HBV Screening - Small group educational session
- Nutrition (Sham Comparator): Small group educational discussion, diet & nutrition resources provided.
  Interventions: Behavioral: Nutrition - Small group educational session

INTERVENTIONS:
Behavioral: HBV Screening - Small group educational session — Small group HBV focused discussion with HBV screening resources.
  Other Names: Hepatitis B screening in Hmong population
  Arms: HBV Screening
Behavioral: Nutrition - Small group educational session — Small group session with diet & nutrition focused, topic related resources provided.
  Other Names: Nutritional education for the Hmong population.
  Arms: Nutrition

SUMMARY:
The purpose of this study is to design an intervention to increase hepatitis B (HBV) screening among Hmong Americans.

DETAILED DESCRIPTION:
The investigators will design an intervention to measure the baseline proportion of Hmong adults (ages 18-64) that have been serologically tested for Hepatitis B. Investigators will work with lay health workers to promote serologically testing for Hepatitis B and increase knowledge of Hepatitis B among Hmong adults. The effectiveness of the lay health worker intervention will be evaluated by conducting a randomized, controlled trial among Hmong adults aged 18-64 not previously tested for hepatitis B.

The primary hypothesis is that the proportion of Hmong adults, ages 18-64 reporting serologically testing for Hepatitis B at post-test will be significantly greater in the intervention group than in the control group.

Secondary hypotheses are:

There will be greater increases in knowledge of Hepatitis B and liver cancer in the intervention group than in the control group.

Participants with greater knowledge of hepatitis B and liver cancer at post-test will be more likely to be serologically tested for hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-64 years
* Hmong ancestry
* Never have been tested for Hepatitis B

Exclusion Criteria:

* Children under the age of 18 years
* Adults over the age of 64 years
* Non-Hmong ancestry
* Previous testing of Hepatitis B

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Obtain HBV Screening Test | September 2006-August 2011

SECONDARY OUTCOMES:
Knowledge and Attitudes Regarding Hepatitis B, Health and Nutrition | September 206 - August 2011

CONTACTS AND LOCATIONS:
Overall Officials: Moon S. Chen, Jr., PhD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Cancer Center, Sacramento, California, United States